CLINICAL TRIAL: NCT04256291
Title: Total Hip Replacement With Ceramic on Ceramic Bearing- Clinical Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807006RINA
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Total Hip Arthroplasty; Total Hip Replacement
Keywords: total hip arthroplasty; ceramic-on-ceramic; total hip replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The pain and severe wear of hip joints caused by osteoarthritis, rheumatoid arthritis, avascular necrosis and trauma can be subjected to total hip replacement (THR). A hip implant consists of 4 components: acetabular cup, femoral stem, articular liner and femoral head. As an ideal material for THR, ceramic possesses excellent biocompatibility and stability in the human bodies. Moreover, ceramic-on-ceramic interface is highly wear-resistant, preventing generation of wear particles. With the development of latest fourth-generation ceramic Delta, larger femoral heads can be manufactured to conform to the size of native femoral heads. The rate of some of the complications after THR, such as dislocation, can be significantly reduced. The purpose of the present study is to carry out a clinical follow up for each patient who has received the ceramic-on-ceramic THR in order to understand the clinical outcome. Furthermore, the possible complications, such as dislocation and squeaking, can be determined.

ELIGIBILITY:
Inclusion criteria:

Patients who has received ceramic-on-ceramic total hip replacement after the year of 2013.

Exclusion criteria:

1. Patients who are unable or unwilling to return for follow-up
2. Patients who have deep periprosthetic joint infection
3. Patients who are diagnosed skeletal dysplasia
4. Patients who suffer from mental disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who has received ceramic-on-ceramic total hip replacement after the year of 2013 at National Taiwan University Hospital Yunlin Branch.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale- Change from baseline at 1 year | Change from baseline at 1 year
  Visual Analogue Scale is a patient-reported outcome measure. The scale ranges from 0 to 10. A score of 0 represents no pain, while a score of 10 represents extreme pain.
Harris Hip Score- Change from baseline at 1 year | Change from baseline at 1 year
  Harris Hip Score includes 4 sections that evaluate pain, function, deformity, and range of motion. Total scores is from 0 to 100, higher scores represent a better outcome.
Oxford Hip Score- Change from baseline at 1 year | Change from baseline at 1 year
  Oxford Hip Score is a patient-reported outcome measure with 12 questions related to the condition of function and pain. Total scores is from 0 to 48, higher scores represent a better outcome.
Radiologic analysis- Change from baseline at 1 year | Change from baseline at 1 year
  Radiologic analysis helps observe the existence of radiolucent lines, which can be analyzed to determine if implant loosening occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Yang-Chen Chou, Study Chair — National Taiwan University Hospital; Chen-Chiang Lin, Study Director — National Taiwan University Hospital
Locations (1):
- Department of Orthopaedics- National Taiwan University Hospital Yunlin Branch, Douliu, Taiwan